CLINICAL TRIAL: NCT05866679
Title: Early Assessment of Ovarian Cancer Aggressiveness by Metabolic Imaging
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspension
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0395; NCI-2023-03931 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hyperpolarized 13-C-pyruvate (Experimental)
  Interventions: Drug: Hyperpolarized 13-C-pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13-C-pyruvate — Given by PO

SUMMARY:
To learn if an MRSI can be performed on a 3T scanner using an investigational contrast drug called hyperpolarized 13-C pyruvate. 3T refers to the "strength" of the MRI machine.

DETAILED DESCRIPTION:
Primary Objective:

1. To assess if increased lactate production measured by HP 13C MRI occurs in suspected ovarian cancer patients who will undergo surgery
2. To evaluate the proportion of increased lactate production in the ovaries measured by HP 13C MRI in low/high ovarian cancer risk patients.

Secondary Objectives:

1. Correlate HP-MR findings to metabolomics, immune profiles, and blood biomarkers of patients undergoing surgical resection.
2. Demonstrate the feasibility and utility of metabolic imaging with HP 13C pyruvate MR in patients with suspected ovarian cancer
3. Correlating imaging findings such as enhancement pattern, ADC values, and advanced image analytics such as texture with pathology and genetic analysis for patients who will undergo surgical resection.

ELIGIBILITY:
Inclusion Criteria:

For the first cohort, the following selection criteria will be applied who are undergoing a screening exam at MD Anderson:

1. Patients with a first degree relative (mother, sister, or daughter) with ovarian cancer or
2. A personal history of breast cancer before age 40 or
3. A personal history of breast cancer diagnosed before age 50, and one or more close relatives diagnosed with breast or ovarian cancer at any age. Two or more close relatives diagnosed with breast cancer before age 50 or with ovarian cancer diagnosed at any age or
4. Ashkenazi Jewish heritage and a personal history of breast cancer before age 50 or
5. Ashkenazi Jewish heritage and a first- or second-degree relative diagnosed with breast cancer before age 50 or with ovarian cancer at any age or
6. Presence of a BRCA1 or BRCA2 mutation or
7. Presence of a mismatch repair gene mutation associated with a hereditary cancer syndrome known as Hereditary Non-Polyposis Colon Cancer (HNPCC)/Lynch syndrome. For the second cohort- 10 Patients will be enrolled who present to MD Anderson for a pelvic ultrasound or have an outside ultrasound or imaging study without a mass or have an adnexal mass (benign) on outside imaging and do not have a high risk for ovarian cancer.

For the third cohort of patients:

10 patients who have suspicion of ovarian malignancy on conventional imaging and will be undergoing surgical resection will be included.

Exclusion Criteria:

(all cohorts)

1. Children, pregnant women, cognitively impaired adults, or prisoners will be excluded from participation.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03 | through study completion: an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Bhosale, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org